CLINICAL TRIAL: NCT03001648
Title: Cumulative Live Birth Rates in Patients With Repeated Implantation Failure (RIF) Undergoing Preimplantation Genetic Screening (PGS )
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Marta Devesa, Staff member of Reproductive Unit, Fundacion Dexeus
Other Study IDs: SMD-DEX-2016-02
Record Dates: First submitted 2016-12-20; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Infertility; Preimplantation Genetic Screening
MeSH Terms: conditions — Infertility | interventions — Phosphatidylglycerols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PGS: Patients with RIF scheduled for PGS (Preimplantation Genetic Screening) with trophectoderm biopsy using arrays comparative genomic hybridation (aCGH) underwent one or more stimulation cycles. If euploid blastocysts were available, patients underwent frozen embryo transfer/s.
  Interventions: Procedure: PGS (Preimplantation Genetic Screening) with trophectoderm biopsy
- Standard IVF: Patients with RIF scheduled for standard IVF (In Vitro Fertilization) underwent a single stimulation cycle with the fresh embryo transfer and the subsequent frozen embryo transfers if there were surplus frozen embryos and the fresh embryo transfer was unsuccessful.

INTERVENTIONS:
Procedure: PGS (Preimplantation Genetic Screening) with trophectoderm biopsy — PGS (Preimplantation Genetic Screening) with trophectoderm biopsy using arrays comparative genomic hybridizatioon (aCGH)
  Groups: PGS

SUMMARY:
This is a single centre retrospective study in repeated implantation failure patients: < 39 years old, at least 4 D3 good quality embryos or 2 good quality blastocysts transferred without implantation, absence of known causes of implantation failures (uterine malformation, thrombophilia, severe male factor, uncontrolled thyroid disfunction, autoimmune disease).

Patients scheduled for PGS underwent one or more stimulation cycles (oocyte or blastocyst banking) in order to maximize chances of embryo transfer. PGS cycles are analyzed globally. Aditionally, PGS cycles with a single stimulation cycle are analyzed in comparison to standard IVF cycles.

ELIGIBILITY:
Inclusion criteria:

* women < 39 years
* repeated implantation failure: at least 4 day 3 good quality embryos or 2 good quality blastocysts transferred without implantation

Exclusion criteria:

* partner with severe male factor, or abnormal sperm Fluorescence in situ hybridization (FISH) analysis
* presence of uni or bilateral hydrosalpinx, uterine malformation, thrombophilia, uncontrolled thyroid disfunction or autoimmune disease

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Repeated implantation failure patients: patients <39 years old that have received at least 4 day 3 good quality embryos or 2 good quality blastocists with no implantation.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cumulative live birth rate | at 24 months of first embryo transfer

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | 6 weeks after embryo transfer
Implantation Rate | 6 weeks after embryo transfer
Miscarriage Rate | Until 20 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona, Barcelona, Spain